CLINICAL TRIAL: NCT00268502
Title: Survey of the Quality of Life of Women
Brief Title: Quality of Life in African-American or Caucasian Female Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IUMC-0209-08B; CDR0000459904 (Registry Identifier: PDQ (Physician Data Query)); IUMC-0502-01B
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer; Cancer Survivor; Depression; Fatigue; Sexual Dysfunction; Sleep Disorders; Spiritual Concerns
Keywords: fatigue; depression; spiritual concerns; sexual dysfunction; sleep disorders; cancer survivor; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Fatigue; Sexual Dysfunction, Physiological; Sleep Wake Disorders | interventions — Therapeutics; Psychiatric Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: study of socioeconomic and demographic variables
Procedure: fatigue assessment and management
Procedure: management of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Studying quality of life in cancer survivors may help determine the long-term effects of breast cancer and may help improve the quality of life for future cancer survivors.

PURPOSE: This clinical trial is studying the quality of life in African-American or Caucasian female breast cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-specific, generic, and global quality of life measures in African-American survivors of breast cancer with Caucasian survivors of breast cancer.
* Compare these quality of life measures in African-American survivors of breast cancer with control group of African-American women with no history of breast cancer.

OUTLINE: Patients and healthy participants complete a battery of quality of life (QOL) questionnaires over approximately 65 minutes by mail or over the phone, including the Sexual Function Index, Functional Assessment of Cancer Therapy - Fatigue, Concerns About Recurrence Scale, and other measures of symptoms/side effects (including sleep problems), the RAND Physical Functioning -10 Scale, Center for Epidemiologic Studies - Depression Scale, assessment of family function/social support, ENRICH Marital Satisfaction Scale, Reed Spiritual Perspective Scale, assessments of coping and body image, Post-Traumatic Growth Inventory, and the Index of Well-being. Demographic, disease, treatment, and comorbidity information, as well as menstrual and gynecological history, work status and insurance history, and a measure of health care provider communication is collected using questionnaires and medical chart review.

PROJECTED ACCRUAL: A total of 195 patients and healthy participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * African-American or Caucasian breast cancer survivor

    * Diagnosed with stage I-III breast cancer between the years of 1995-2003
    * Receiving follow up care at the Indiana University Cancer Center (IUCC), the IUCC Northside Clinic, Spring Mill Clinic, or Wishard Memorial Hospital
  * Healthy African-American

    * Acquaintance of an African-American breast cancer survivor
    * Not known to have breast cancer

PATIENT CHARACTERISTICS:

* Female

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Russell, RN, DNS, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States